CLINICAL TRIAL: NCT02864628
Title: A Partially Randomized, Partly Placebo Controlled Phase I Trial to Evaluate the Safety, Tolerability and Immunogenicity of the Recombinant MVA-BN® RSV Vaccine After Intranasal and Intramuscular Administration
Brief Title: RSV-MVA-BN Vaccine Phase I Trial, Intranasal Application in Adults.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Protocol was withdrawn from IND
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RSV-MVA-006
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: RSV Vaccines; Respiratory Syncytial Virus Vaccines
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1 (Experimental): ≥55 year old healthy subjects, receiving either 5x10E7 TCID50 MVA-BN-RSV or Placebo intranasal application
  Interventions: Biological: MVA-BN-RSV; Other: Placebo
- Group 2 (Experimental): ≥55 year old healthy subjects, receiving either 1x10E8 TCID50 MVA-BN-RSV or Placebo intranasal application
  Interventions: Biological: MVA-BN-RSV; Other: Placebo
- Group 3 (Experimental): ≥55 year old healthy subjects, receiving either 5x10E8 TCID50 MVA-BN-RSV or Placebo intranasal application
  Interventions: Biological: MVA-BN-RSV; Other: Placebo
- Group 4 (Experimental): ≥55 year old healthy subjects, receiving 5x10E8 TCID50 MVA-BN-RSV intranasal and intramuscular application
  Interventions: Biological: MVA-BN-RSV
- Group 5 (Experimental): ≥55 year old healthy subjects, receiving 5x10E8 TCID50 MVA-BN-RSV intramuscular application
  Interventions: Biological: MVA-BN-RSV

INTERVENTIONS:
Biological: MVA-BN-RSV — MVA-mBN294B
Other: Placebo — Tris Buffered Saline
  Arms: Group 1; Group 2; Group 3

SUMMARY:
A total of 96 subjects will be recruited into 5 groups. Each subject will receive either two vaccinations with MVA-BN-RSV vaccine or placebo.

ELIGIBILITY:
Inclusion Criteria:

* signed and dated an informed consent form and HIPAA.
* Subjects without symptomatic cardiopulmonary and/or metabolic disease.
* Body mass index (BMI) ≥ 18.5 and ≤ 34.9.
* Negative human immunodeficiency virus antibody test (anti-HIV), HBsAG and HCV virus.
* Electrocardiogram (ECG) without clinically significant acute findings.
* WOCBP must have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to each vaccination.

Exclusion Criteria:

* History of nasal or sinus surgery within six months prior to screening or planned nasal or sinus surgery during the trial
* Active or recent history (within 6 months prior to screening) of chronic sinusitis, nasopharyngeal abnormalities and/or symptoms such as polyps or deviated septum
* pregnant or breast-feeding women.
* History or current clinical manifestation of any serious medical condition.
* History of or active autoimmune disease.
* Known or suspected impairment of immunologic functions including, but not limited to chronic inflammatory bowel disorders, diabetes mellitus type I.
* Knowledge/history of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* History of anaphylaxis or severe allergic reaction to any vaccine.
* Chronic systemic administration defined as more than 14 days of > 5 mg prednisone per day

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09 (Estimated); Primary Completion 2017-10-27 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
Occurrence of serious adverse events | Screening up to week 34 after first vaccination
  Occurrence, relationship to the trial vaccine and intensity of any serious adverse event (SAE).

SECONDARY OUTCOMES:
RSV-specific humoral immune response | humoral immune response is measured up to week 34
  To assess the RSV-specific serum antibody responses

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Fierro, MD, Principal Investigator — Johnson County Clin-Trials (JCCT)

IPD SHARING:
Plan to Share IPD: Undecided